CLINICAL TRIAL: NCT03857204
Title: Fetus Weight Estimation by Ultrasound Data Collection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0108-18-HYMC
Record Dates: First submitted 2019-02-12; First posted 2019-02-27 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Fetal Weight
MeSH Terms: conditions — Fetal Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- performing US scans for fetal weight assessment. (Experimental)
  Interventions: Device: SAMPL plain wave algorithm

INTERVENTIONS:
Device: SAMPL plain wave algorithm — SAMPL's plain-wave algorithm allowing portable US or Wireless Probe scanning - thus enabling clinicians with more flexible point-of-care locations when performing US scans for fetal weight assessment.

SUMMARY:
This research aims to allow deployment & optimization of SAMPL plain wave algorithm so as to make required advancement towards a light-weight portable US platform or wireless probe - thus elevating clinician's care level and patient treatment by allowing more scan availability and flexibility.

ELIGIBILITY:
Inclusion Criteria:

1. Women between 24+0 weeks and 41+6 weeks gestation.
2. Women with a singleton viable pregnancy.

Exclusion Criteria:

None

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
US scans for fetal weight assessment | 1 year
  1) To evaluate SAMPL's plain-wave algorithm allowing portable US or Wireless Probe scanning - thus enabling clinicians with more flexible point-of-care locations when performing US scans for fetal weight assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Alon Shrim, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hille Yaffe Medical Center, Hadera, Israel